CLINICAL TRIAL: NCT04848974
Title: Phase Ib/II Study of Uproleselan Added to Cladribine Plus Low Dose Cytarabine (LDAC) Induction Followed by Consolidation With Uproleselan Plus Cladribine Plus LDAC in Patients With Treated Secondary AML (TS-AML)
Brief Title: Uproleselan, Cladribine, and Low Dose Cytarabine for the Treatment of Patients With Treated Secondary Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0988; NCI-2021-02298 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0988 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-05; First posted 2021-04-19 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Secondary Acute Myeloid Leukemia
MeSH Terms: interventions — Cladribine; Cytarabine; uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 (Experimental): INDUCTION THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine SC BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.
  CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV QD on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Uproleselan
- Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (Experimental): INDUCTION THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine SC BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.
  CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV QD on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Uproleselan
- Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (Experimental): INDUCTION THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine SC BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.
  CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV QD on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Uproleselan

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Uproleselan — Given IV
  Other Names: GMI-1271

SUMMARY:
This phase Ib/II trial finds out the best dose and effect of cladribine and low dose cytarabine when given in combination with uproleselan in treating patients with treated secondary acute myeloid leukemia. Chemotherapy drugs, such as uproleselan, cladribine, and low dose cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability, and recommended phase II dose (RP2D) of uproleselan combined with cladribine + low dose cytarabine (LDAC) in patients with treated-secondary acute myeloid leukemia (AML) (ts-AML).

SECONDARY OBJECTIVES:

I. To assess the efficacy (overall response rate [ORR], complete response [CR], complete response without blood count recovery [CRi], CR with partial hematologic recovery [CRh], partial response [PR], or morphologic leukemia-free state of uproleselan combined with cladribine + LDAC in patients with ts-AML.

II. To assess the rate of minimal residual disease (MRD) negativity by flow cytometry at response.

III. To assess overall survival (OS), remission duration (CRd), and progression-free survival (PFS) in patients with ts-AML treated with uproleselan combined with cladribine + LDAC.

IV. To assess the rate of complete cytogenetic response (CCyR) in patients with ts-AML with abnormal baseline karyotype, treated with uproleselan combined with cladribine + LDAC.

V. To assess toxicity and induction mortality of patients with AML treated with uproleselan added to cladribine + LDAC.

EXPLORATORY OBJECTIVES:

I. To explore biomarkers of response and resistance in patients with ts-AML treated with uproleselan combined with cladribine + LDAC.

II. To examine the correlation of E-selectin ligand-forming glycosylation genes of leukemic blasts with clinical outcome.

OUTLINE: This is a phase I, dose-escalation study of cladribine and cytarabine followed by a phase II study.

INDUCTION THERAPY: Patients receive uproleselan intravenously (IV) over 20 minutes on day 1 and every (Q) 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine subcutaneously (SC) twice daily (BID) on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.

CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV once daily (QD) on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of treated secondary-AML (TS-AML) who have not received therapy for their AML will be eligible.
2. TS-AML is defined as AML arising from a previously treated antecedent myeloid neoplasm (myelodysplastic syndrome or myeloproliferative neoplasm that has been previously treated with hypomethylating agents).
3. Patients must be at least 7 days from their last therapy for the antecedent myeloid neoplasm
4. Age >/= 18 years.
5. Adequate organ function as defined below:

   * liver function (total bilirubin < 2mg/dL, AST and/or ALT <3 x ULN - or <5 x ULN if related to leukemic involvement)
   * kidney function (creatinine < 1.5 x ULN ).
   * known cardiac ejection fraction of > or = 45% within the past 6 months
6. ECOG performance status of ≤ 2.
7. A negative urine or serum pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
8. Patient must have the ability to understand the requirements of the study and informed consent. A signed informed consent by the patient is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with documented hypersensitivity to any of the components of the chemotherapy program.
4. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
5. Prior treatment with uproleselan.
6. Patients with a diagnosis of acute promyelocytic leukemia (AML-M3) will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2; Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2; Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2: INDUCTION THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine SC BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.
  CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV QD on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given SC
  Uproleselan: Given IV
Period: Overall Study
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Started | 3 | 9 | 25
Completed | 3 | 9 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Total
Number analyzed (Participants) | 3 | 9 | 25 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 2 | 7 | 23 | 32
Age, Continuous [Median (Full Range); unit: years] | 76 [58 to 80] | 68 [59 to 77] | 73 [61 to 86] | 73 [58 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 19 | 24
  Male | 2 | 5 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 3 | 6 | 24 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 25 | 37

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose
Description: During safety lead-in, we will use the Bayesian optimal interval (BOIN) design to identify the RP2D of the combination therapy. If the observed DLT rate at the current dose is . 0.236, escalate the dose to the next higher dose level;
  . if the observed DLT rate at the current dose is . 0.359, de-escalate the dose to the next lower dose level; otherwise, stay at the current dose.
Time Frame: Up to two courses of Induction therapy, each course is approximately 4 weeks +/- 7 days
Measure: Number; unit: mg/m^2
Groups:
- All Participants Enrolled in Phase 1b: INDUCTION THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q 12 hours on days 2-12, cladribine IV over 1-2 hours on days 1-5 and cytarabine SC BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle.
  CONSOLIDATION/MAINTENANCE THERAPY: Patients receive uproleselan IV over 20 minutes on day 1 and Q12 hours on days 2-1. Patients who have achieved at least CR/CRi or morphologic leukemia-free state after induction therapy receive uproleselan IV QD on days 1-12. Patients also receive cladribine IV over 1-2 hours on days 1-3 and cytarabine SC BID on days 1-10. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given SC
  Uproleselan: Given IV
Arm/Group | All Participants Enrolled in Phase 1b
Number analyzed (Participants) | 12
mg/m^2 | 5

2. Secondary Outcome: Number of Participants With a Response
Description: Response is Complete Remission (CR) + Complete Remission Without Count Recovery (CRi) + Morphologic Leukemia-Free State (MLFS) - CR is Disappearance of all clinical and/or radiologic evidence of disease, including extramedullary leukemia. Neutrophil count . 1.0 x 10^9/L and platelet count . 100 x 10^9/L, and bone marrow differential showing . 5% blasts. CRi is Have met all criteria for CR, except for either residual neutropenia (ANC < 1.0 x 10^9/L) or thrombocytopenia (platelet count < 100 x 10^9/L). MLFS is Bone marrow differential showing < 5% blasts, no evidence of peripheral blasts or extramedullary disease, but without peripheral blood count recovery to neutrophil count . 1.0 x 10^9/L & platelet count . 100 x 10^9/L.
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Participants | 1 | 4 | 9

3. Secondary Outcome: Number of Participants With Complete Response (CR)
Description: Disappearance of all clinical and/or radiologic evidence of disease, including extramedullary leukemia. Neutrophil count . 1.0 x 10^9/L and platelet count . 100 x 10^9/L, and bone marrow differential showing . 5% blasts.
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Participants | 0 | 2 | 2

4. Secondary Outcome: Number of Participants With Complete Remission Without Blood Count Recovery (CRi)
Description: Have met all criteria for CR, except for either residual neutropenia (ANC < 1.0 x 10^9/L) or thrombocytopenia (platelet count < 100 x 10^9/L).
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Participants | 0 | 1 | 5

5. Secondary Outcome: Number of Participants to Reach Morphologic Leukemia-free State (MLFS)
Description: Bone marrow differential showing < 5% blasts, no evidence of peripheral blasts or extramedullary disease, but without peripheral blood count recovery to neutrophil count . 1.0 x 10^9/L & platelet count . 100 x 10^9/L.
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Participants | 1 | 1 | 2

6. Secondary Outcome: Number of Minimal Residual Disease (MRD) Negativity in Responders
Description: Measures the Minimal Residual Disease (MRD) negativity in participants who achieve Complete Remission (CR) or Complete remission without count recovery (CRi) - CR is Disappearance of all clinical and/or radiologic evidence of disease, including extramedullary leukemia. Neutrophil count . 1.0 x 10^9/L and platelet count . 100 x 10^9/L, and bone marrow differential showing . 5% blasts. CRi is Have met all criteria for CR, except for either residual neutropenia (ANC < 1.0 x 10^9/L) or thrombocytopenia (platelet count < 100 x 10^9/L).
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 1 | 4 | 7
Participants | 1 | 2 | 2

7. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause.
Time Frame: From treatment start to the date of death or last follow-up, whichever occurred first, Up to 3 years, 4 months and 14 days
Measure: Median (Full Range); unit: Months
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Months | 0.8 [0.6 to 4.8] | 5.5 [1.7 to 26.3] | 3.8 [0.4 to 12.7]

8. Secondary Outcome: Complete Remission Duration
Description: The date of Complete Response to the date of loss of response or last follow-up.
Time Frame: From date of CR/CRi to date of disease relapse, death or last follow-up, whichever occurred first, assessed up to 4.5 years
Reporting Status: Not Posted

9. Secondary Outcome: Event-free Survival
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: From treatment start to date of death, relapse or last follow-up, whichever occurred first, Up to 3 years, 4 months and 14 days
Measure: Median (Full Range); unit: Months
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Months | 0.6 [0.5 to 2.8] | 3.1 [0.7 to 26.3] | 1.7 [0.4 to 7.2]

10. Secondary Outcome: The Number of Participants With Complete Cytogenetic Response (CCyR)
Description: To assess the rate of complete cytogenetic response (CCyR) in patients with abnormal baseline karyotype, treated with uproleselan combined with cladribine + LDAC. Participants were evaluated for abnormal baseline karyotype and evaluated again after treatment.
Time Frame: Up to 3 years, 4 months and 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 1 | 2 | 5
Participants | 1 | 1 | 2

11. Secondary Outcome: Induction Mortality, Number of Participants
Description: Number of participants who died during the induction period of therapy.
Time Frame: Up to two courses of Induction therapy, each course is approximately 4 weeks +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
Number analyzed (Participants) | 3 | 9 | 25
Participants | 0 | 0 | 4

ADVERSE EVENTS:
Time Frame: From treatment start to the date of death or last follow-up, whichever occurred first, Up to 3 years, 4 months and 14 days
Arm/Group | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/3 | 7/9 | 24/25
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/9 | 15/25
Other Adverse Events (participants affected / at risk) | 3/3 | 6/9 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 (N=3) | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (N=9) | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (N=25)
Chills (General disorders) | 0 (0) | 0 (0) | 1/15 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1/15 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0/15 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1 Treatment Dose Level -1 Cladaribine 3.75mg/m^2 (N=3) | Ph 1 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (N=9) | Ph 2 Treatment Dose Level 1 Cladaribine 5 mg/m^2 (N=25)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Bleeding gums (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Redness sacrum (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Sacral wound (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
streptococcus (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Infection-Other (Specify) (Infections and infestations) | 3 (5) | 3 (7) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4)
hypervolemia (General disorders) | 0 (0) | 0 (0) | 3 (4)
tachypnea (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Weight loss (Investigations) | 0 (0) | 0 (0) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Back pain (General disorders) | 0 (0) | 0 (0) | 4 (5)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Lethargy (General disorders) | 0 (0) | 0 (0) | 5 (5)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain (General disorders) | 0 (0) | 0 (0) | 7 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7)
Pain (General disorders) | 0 (0) | 0 (0) | 5 (9)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (10)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 7 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 10 (12)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 11 (13)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 11 (14)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 9 (20)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhagic Cystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC--Select (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT04848974/Prot_SAP_001.pdf